CLINICAL TRIAL: NCT03121690
Title: The Applicability of Different Scoring Systems and Use of Steroids in the Treatment of Hospital Acquired Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rabab Hamed Hassan, specialist of chest and tuberculosis, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17200051
Record Dates: First submitted 2017-04-10; First posted 2017-04-20 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Pneumonia Hospital Acquired
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- prednisone (Experimental): prednisone 40 mg/day for 7 days
  Interventions: Drug: Prednisone; Drug: placebo
- placebo (Experimental): 5ml saline /day for 7 days
  Interventions: Drug: Prednisone; Drug: placebo

INTERVENTIONS:
Drug: Prednisone — prednisone 40 mg/day for 7 days
  Other Names: hostacortin
Drug: placebo — 5ml saline / day for 7 days

SUMMARY:
Cross sectional randomized clinical trial study will be done at Respiratory intensive care unit and Chest department at Assiut University Hospitals on All patients who developed hospital acquired pneumonia including ventilator associated pneumonia through two years duration to assess the prognostic value of different severity scores including (PSI, CURB65, SMART COP, IDSA/ATS and SOAR) in patients with HAP, assess platelet count as a marker for severity, evaluate efficacy and safety of adjuvant systemic steroids in patients with severe conditions and measurement of cortisol level to assess steroid response before administration.

DETAILED DESCRIPTION:
The following parameters will be recorded:

* Demographic data: including age, sex, smoking history.
* Clinical data: Glasgow coma scales, Co-morbidities are determined by reviewing the patients' clinical histories, chest examination.
* Vital signs: including body temperature, respiratory rate, heart rate, and arterial blood pressure.
* Oxygenation data: including arterial blood gases in fixed days (at the start, 3rd day and 7th day of steroid administration), ratio of partial oxygen tension in arterial blood to fraction of inspired oxygen (PaO2/FiO2 ratio).
* Laboratory data include complete blood picture focusing on leukocytic count and platelets, kidney and liver function tests, serum electrolytes, Erythrocyte sedimentation rate, C reactive protein, sputum culture and cortisol level before steroid administration.
* Radiology data include chest X-ray and chest ultrasonography at the day of diagnosis and at 7th day of steroid administration. Chest CT will be done if possible.

Procedures: Systemic steroids will be administered early with a dosages equivalent to prednisone 40 mg/day for 7 days which is considered as a "stress dose" of systemic corticosteroids for pneumonia. The patients will also receive the appropriate initial intravenous antibiotic medication and the standard care as recommended in RICU policy. Cortisol level will be measured before steroid administration.

ELIGIBILITY:
Inclusion Criteria:

This study will be conducted on admitted patients aged ≥18 years that developed hospital acquired pneumonia including ventilator associated pneumonia. Its diagnosis is confirmed by developing pneumonia after 48 H of admission and they had new or progressive infiltrates on the chest X-ray with one of the 3 requirements of: fever more than 37.8 C or purulent sputum or leukocytosis.

Exclusion Criteria:

1. Patients having lung cancer and those who hadn't the full data for scoring fulfilled.
2. Chronically immunosuppressed patients (chemotherapy, human immunodeficiency virus infection, or other immunosuppressive agents).
3. Condition requiring prolonged steroid use > 0.5 mg/kg/day of prednisone equivalent.
4. Major gastrointestinal bleeding within 3 months.
5. Patients with prolonged intubation and having tracheostomy.
6. Patients with neurological disorders or encephalopathy.
7. Patients with pandemic H1N1 influenza A pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Hospital mortality | 28 days
  measure the predicting 28 day mortality for all included cases.

SECONDARY OUTCOMES:
Percentage of ICU needing | 28 days
  the need of non-invasive ventilation and mechanical ventilation
Time to clinical stability | 28 days
  measure time to resolution of vital signs, ability to eat and mental status
complications of hospitalization | 28 days
  occurrence of complication arising during hospitalization (ARDS, shock, sepsis, major arrhythmia include atrial fibrillation and supraventricular tachycardia , renal failure, electrolyte disturbance, deep venous thrombosis and GIT bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abd-Elatif bayoumi, lecturer, Principal Investigator — Assiut University
Locations (1):
- Rabab Hamed Hassan, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided